CLINICAL TRIAL: NCT00887484
Title: A Single-blind, Randomized, Comparative Pilot Study Evaluating the Tolerability of Two Topical Combination Therapies in the Treatment of Acne Vulgaris
Brief Title: A Comparative Study of the Tolerability of Two Combination Therapies for the Treatment of Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114544
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Acne Vulgaris
Keywords: Acne; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate benzoyl peroxide combination; Benzoyl Peroxide; Adapalene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clindoxyl Gel (Experimental): Subject will apply both study products in a split-face fashion. Study products will be applied once-daily in the evening.
  Interventions: Drug: BENZOYL PEROXIDE/ CLINDAMYCIN
- Epiduo gel (Active Comparator): Subject will apply both study products in a split-face fashion. Study products will be applied once-daily in the evening.
  Interventions: Drug: BENZOYL PEROXIDE/ ADAPALENE

INTERVENTIONS:
Drug: BENZOYL PEROXIDE/ CLINDAMYCIN — Commencing at baseline, subjects will apply once daily both treatment arm #1 and treatment arm #2 in a bilateral split-face fashion (allocation to left and right side randomly assigned) for an initial 2 weeks. At 2 weeks, subjects will apply benzoyl peroxide/clindamycin gel to the entire face for an additional 6 weeks.
  Arms: Clindoxyl Gel
Drug: BENZOYL PEROXIDE/ ADAPALENE — Commencing at baseline, subjects will apply once daily both treatment arm #1 and treatment arm #2 in a bilateral split-face fashion (allocation to left and right side randomly assigned) for an initial 2 weeks. At 2 weeks, subjects will apply benzoyl peroxide/clindamycin gel to the entire face for an additional 6 weeks.
  Arms: Epiduo gel

SUMMARY:
The purpose of this study is to compare the tolerability of topical combination therapies in the treatment of facial acne.

DETAILED DESCRIPTION:
The purpose of this study is to compare the tolerability of topical combination therapies in the treatment of facial acne.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 21 years of age, in good general health with documented diagnosis of acne vulgaris.
* Female subjects of childbearing potential must have a negative pregnancy test. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception Abstinence is considered an acceptable method of contraception.
* Inflammatory (papules and pustules) and non-inflammatory (open and closed comedones) facial lesions.
* The ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study
* Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed

Exclusion Criteria:

* Female subjects who are pregnant, trying to become pregnant or breastfeeding.
* Subjects who have any clinically relevant finding at their baseline physical other than acne vulgaris.
* History or presence of regional enteritis or inflammatory bowel disease (eg, ulcerative colitis, pseudomembranous colitis, chronic diarrhea, or a history of antibiotic-associated colitis) or similar symptoms.
* Use of topical antibiotics or anti-acne medications on the face and systemic antibiotics within the past 2 and 4 weeks, respectively.
* Use of topical corticosteroids on the face or systemic corticosteroids within the past 4 weeks. Use of inhaled, intra-articular or intra-lesional (other than for facial acne lesions) steroids is acceptable.
* Use of systemic retinoids within the past 6 months.
* Facial procedures performed by an esthetician, beautician, physician, nurse, or other practitioner, within the past 4 weeks or during the conduct of the study.
* Known hypersensitivity or previous allergic reaction to any of the active components, lincomycin, adapalene, clindamycin, benzoyl peroxide or excipients of the study product.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Argentina (4):
  - Centro de Investigación y Prevencion de Enfermidades Cardiovasculares, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - LUMIPIEL - Centro Dermatológico, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Buenos Aires Skin, Ciudad de Buenos Aires, Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 114544 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114544 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114544 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114544 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114544 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical research center
Groups:
- Clindoxyl and Epiduo Gels: Commencing at baseline, participants will apply clindoxyl and epiduo gels once daily in a bilateral split-face fashion (Split Face Treatment Period; allocation to left and right side randomly assigned) for an initial 2 weeks. At Week 5, during the Full Face Treatment Period, participants will apply clindoxyl gel to the entire face for an additional 4 weeks.
Period: Split Face Treatment (Weeks 1 and 2)
Arm/Group | Clindoxyl and Epiduo Gels
Started | 48
Completed | 48
Not Completed | 0
Period: Full Face Treatment (Weeks 5 and 8)
Arm/Group | Clindoxyl and Epiduo Gels
Started | 48
Completed | 45
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clindoxyl and Epiduo Gels
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (5.5)
Gender [Count of Participants; unit: Participants]
  Female | 10
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 48
Investigators Static Global Assessment (ISGA) [Number; unit: Participants] — The investigator rated the participants' skin using the 6-point ISGA: 0=clear, clear skin with no inflammatory lesions (ILs) or non-ILs; 1=almost clear, rare non-ILs with no more than one small IL; 2=mild, some non-ILs with no more than a few ILs (papules/pustules only, no nodular lesions [NLs]); 3=moderate, up to many non-ILs and may have some ILs, but no more than one small NL; 4=severe, up to many non-IL and ILs, but no more than a few NLs; 5=many non-IL and ILs and more than a few NLs. May have cystic lesions. Participants with grades of 2-4 were eligible for enrollment in this study.
  Participants
    Mild | 14
    Moderate | 31
    Severe | 3
Inflammatory Acne Lesion Count [Mean (Standard Deviation); unit: Inflammatory lesions] — Inflammatory acne lesion count at baseline (number of pustules and papules).
  Inflammatory lesions | 14.2 (9.1)
Non-Inflammatory Acne Lesion Count [Mean (Standard Deviation); unit: Non-Infammatory acne lesions] — Non-Inflammatory acne lesion count at baseline (number of whiteheads and blackheads)
  Non-Infammatory acne lesions | 24.8 (12.8)
Total Acne Lesion Count [Mean (Standard Deviation); unit: Acne lesions] — Total acne lesion count (includes inflammatory and non-inflammatory lesions)
  Acne lesions | 39.1 (13.0)

OUTCOME MEASURES:

1. Primary Outcome: Erythema (Redness)
Description: Signs and symptoms of tolerability (erythema, peeling, dryness, and irritant/allergic contact dermatitis)on the face.
  Erythema, peeling, dryness, and irritant/allergic contact dermatitis were graded using the following scale: 0, None; 1, Slight; 2, Moderate; 3, Intense.
Time Frame: Weeks 1 and 2
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Clindoxyl Gel: Clindoxyl gel was applied to one side of the face in a randomized fashion. This study product was applied once-daily in the evening.
- Epiduo Gel: Epiduo gel was applied to one side of the face in a randomized fashion. This study product was applied once-daily in the evening.
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
units on a scale
  Week 1 | 0.66 (0.70) | 0.91 (0.78)
  Week 2 | 0.55 (0.62) | 0.74 (0.64)

2. Secondary Outcome: Erythema (Redness)
Description: as for outcome 1
Time Frame: Weeks 5 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Clindoxyl Gel: Subjects applied Clindoxyl gel to their entire face once-daily in the evening.
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
units on a scale
  Week 5 | 0.22 (0.42)
  Week 8 | 0.19 (0.50)

3. Secondary Outcome: Skin Dryness
Description: as for outcome 1
Time Frame: Weeks 5 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
units on a scale
  Week 5 | 0.20 (0.46)
  Week 8 | 0.04 (0.29)

4. Primary Outcome: Skin Dryness
Description: as for outcome 1
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
units on a scale
  Week 1 | 0.47 (0.55) | 0.96 (0.75)
  Week 2 | 0.40 (0.58) | 0.64 (0.74)

5. Primary Outcome: Skin Peeling
Description: Signs and symptoms of tolerability (erythema, peeling, dryness, and irritant/allergic contact dermatitis)on the face.
  Erythema, peeling, dryness, and irritant/allergic contact dermatitis were graded using the following scale: 0, None; 1, Slight; 2, Moderate; 3,Intense.
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Epiduo: Epiduo gel was applied to one side of the face in a randomized fashion. This study product was applied once-daily in the evening.
Arm/Group | Clindoxyl Gel | Epiduo
Number analyzed (Participants) | 48 | 48
units on a scale
  Week 1 | 0.34 (0.52) | 0.68 (0.78)
  Week 2 | 0.40 (0.61) | 0.60 (0.68)

6. Primary Outcome: Irritant/Allergic Contact Dermatitis
Description: as for outcome 1
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
units on a scale
  Week 1 | 0.04 (0.20) | 0.04 (0.20)
  Week 2 | 0.04 (0.20) | 0.04 (0.20)

7. Secondary Outcome: Skin Peeling
Description: as for outcome 1
Time Frame: Weeks 5 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
units on a scale
  Week 5 | 0.13 (0.40)
  Week 8 | 0.06 (0.25)

8. Secondary Outcome: Irritant/Allergic Contact Dermatitis
Description: as for outcome 1
Time Frame: Weeks 5 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
units on a scale
  Week 5 | 0.00 (0.00)
  Week 8 | 0.00 (0.00)

9. Secondary Outcome: Investigators Static Global Assessment
Description: ISGA is evaluated using the following scale: 0, Clear: Clear skin with no lesions; 1, Almost Clear: Rare non-inflammatory lesions; 2, Mild: Some non-inflammatory lesions with no more than a few inflammatory lesions but no nodular lesions); 3, Moderate: Up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than 1 small nodular lesion; 4, Severe: Up to many non-inflammatory and inflammatory lesions, but no more than a few nodular lesions; 5, Very Severe: Many non-inflammatory and inflammatory lesions and more than a few nodular lesions. May have cystic lesions.
Time Frame: Baseline, Weeks 5, 8
Population: For the first 2 weeks, participants apply one of the drugs (Clindoxyl or Epiduo) to one side of the face and the other drug to the other side of their face. After week 2, participants apply Clindoxyl to their entire face and do not use Epiduo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
units on a scale
  Baseline | 2.77 (0.56)
  Week 5 | 1.89 (0.75)
  Week 8 | 1.62 (0.92)

10. Secondary Outcome: Total Acne Lesion Counts
Description: Total acne lesion counts - includes both inflammatory acne lesions (pustules, papules), noninflammatory lesions (whiteheads and blackheads),
Time Frame: Baseline, Weeks 5 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Acne Lesions
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Acne Lesions
  Baseline | 39.06 (12.95)
  Week 5 | 15.96 (10.37)
  Week 8 | 13.77 (11.50)

11. Secondary Outcome: Inflammatory Acne Lesion Counts
Description: Total number of inflammatory acne lesions (pustules, papules) at each timepoint.
Time Frame: Baseline, Weeks 5 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Acne Lesions
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Acne Lesions
  Baseline | 14.23 (9.06)
  Week 5 | 4.60 (3.93)
  Week 8 | 4.26 (5.84)

12. Secondary Outcome: Non-inflammatory Acne Lesion Counts
Description: Total number of non-inflammatory acne lesions (whiteheads and blackheads) at each timepoint.
Time Frame: Baseline, Weeks 5 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Acne Lesions
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Acne Lesions
  Baseline | 24.83 (12.84)
  Week 5 | 11.36 (7.89)
  Week 8 | 9.51 (8.53)

13. Secondary Outcome: Skindex-29 Quality of Life Questionnaire (QoL) - Symptomatic Domain
Description: Skindex-29 is a self-administered (by participants at each time point) QoL questionnaire comprised of 29 items (it.) scored on a 5-point scale (0=never, 1=rarely, 2=sometimes, 3=often, 4=all the time) covering 3 domains: emotional (10 it.); symptomatic (7 it.); functional (12 it.). Domain scores range from 0 to 40, 0 to 28, and 0 to 48, respectively. Lower scores=better QoL. The symptomatic score (score=0 to 28)=(sum of the 7 individual item scores) * 100/28.
Time Frame: Baseline, Weeks 2 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale
  Baseline | 20.91 (15.73)
  Week 2 | 21.58 (14.17)
  Week 8 | 13.75 (14.03)

14. Secondary Outcome: Quality of Life Questionnaire - Emotional Domain
Description: Skindex-29 is a self-administered (by participants at each time point) QoL questionnaire comprised of 29 items (it.) scored on a 5-point scale (0=never, 1=rarely, 2=sometimes, 3=often, 4=all the time) covering 3 domains: emotional (10 it.); symptomatic (7 it.); functional (12 it.). Domain scores range from 0 to 40, 0 to 28, and 0 to 48, respectively. Lower scores=better QoL. The emotional score (score=0 to 40)=(sum of the 10 individual item scores) * 100/40.
Time Frame: Baseline, Weeks 2 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale
  Baseline | 25.32 (19.73)
  Week 2 | 19.38 (18.68)
  Week 8 | 16.42 (19.08)

15. Secondary Outcome: Quality of Life Questionnaire - Functional Domain
Description: Skindex-29 is a self-administered (by participants at each time point) QoL questionnaire comprised of 29 items (it.) scored on a 5-point scale (0=never, 1=rarely, 2=sometimes, 3=often, 4=all the time) covering 3 domains: emotional (10 it.); symptomatic (7 it.); functional (12 it.). Domain scores range from 0 to 40, 0 to 28, and 0 to 48, respectively. Lower scores=better QoL. The functional score (score=0 to 48)=(sum of the 12 individual item scores) * 100/48.
Time Frame: Baseline, Weeks 2 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale
  Baseline | 8.59 (13.98)
  Week 2 | 6.30 (11.77)
  Week 8 | 5.19 (11.78)

16. Secondary Outcome: Quality of Life Questionnaire - Global Score
Description: Skindex-29 is a self-administered (by participants at each time point) QoL questionnaire comprised of 29 items (it.) scored on a 5-point scale (0=never, 1=rarely, 2=sometimes, 3=often, 4=all the time) covering 3 domains: emotional (10 it.); symptomatic (7 it.); functional (12 it.). Domain scores range from 0 to 40, 0 to 28, and 0 to 48, respectively. Lower scores=better QoL. A Global Score (range 0-100)=(sum of all 29 individual item scores) * 100/116.
Time Frame: Baseline, Weeks 2 and 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale
  Baseline | 8.59 (13.98)
  Week 2 | 6.30 (11.77)
  Week 8 | 5.19 (11.78)

17. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Redness at Weeks 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint using the following scale: 0, None; 1, Very minimal; 2, Mild; 3, Moderate; 4, Severe.
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 1.09 (1.18) | 1.72 (1.21)
  Week 2 | 0.72 (0.86) | 1.15 (1.07)

18. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Redness at Week 8
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 0, None; 1, Very minimal; 2, Mild; 3, Moderate; 4, Severe.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 0.77 (1.09)

19. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Dryness at Weeks 1 and 2
Description: as for outcome 17
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 1.30 (1.14) | 1.81 (1.14)
  Week 2 | 1.00 (0.87) | 1.41 (1.17)

20. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Dryness at Week 8
Description: as for outcome 18
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 0.64 (0.97)

21. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Burning at Weeks 1 and 2
Description: as for outcome 17
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 0.91 (1.23) | 1.68 (1.20)
  Week 2 | 0.72 (0.89) | 1.30 (1.23)

22. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Burning at Week 8
Description: as for outcome 18
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 0.36 (0.76)

23. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Itching at Weeks 1 and 2
Description: as for outcome 17
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 0.64 (1.11) | 1.02 (1.34)
  Week 2 | 0.72 (0.96) | 0.93 (1.00)

24. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Itching at Week 8
Description: as for outcome 18
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 0.26 (0.49)

25. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Scaling at Weeks 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint using the following scale: 0, None; 1, Very minimal; 2, Mild; 3, Moderate; 4, Severe; 5, Very Severe.
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 0.79 (1.18) | 1.43 (1.41)
  Week 2 | 0.59 (0.69) | 1.04 (1.07)

26. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Scaling at Week 8
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 0, None; 1, Very minimal; 2, Mild; 3, Moderate; 4, Severe; 5, Very Severe.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 0.45 (0.83)

27. Secondary Outcome: Product Acceptability and Preference Questionnaire - Ease of Application of Product at Weeks 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint using the following scale: 1, Very easy; 2, Easy; 3, Neutral; 4, Difficult.
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 1.30 (0.51) | 1.32 (0.56)
  Week 2 | 1.35 (0.53) | 1.39 (0.61)

28. Secondary Outcome: Product Acceptability and Preference Questionnaire - Ease of Application of Product at Week 8
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 1, Very easy; 2, Easy; 3, Neutral; 4, Difficult.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 1.26 (0.44)

29. Secondary Outcome: Product Acceptability and Preference Questionnaire - Comfort of Skin at Weeks 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint using the following scale: 1, Very Comfortable; 2, Comfortable; 3, Somewhat Comfortable; 4, Somewhat Uncomfortable; 5, Uncomfortable.
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 2.81 (0.88) | 3.15 (1.08)
  Week 2 | 2.39 (0.93) | 2.67 (0.94)

30. Secondary Outcome: Product Acceptability and Preference Questionnaire - Comfort of Skin at Week 8
Description: as for outcome 29
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 1.83 (0.92)

31. Secondary Outcome: Product Acceptability and Preference Questionnaire - Which Study Product is Subject More Satisfied With? at Weeks 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint using the following choices: Epiduo, Clindoxyl Gel, Both Treatments Equally.
Time Frame: Weeks 1 and 2
Population: ITT. Data are presented for only those participants completing the questionnaire.
Measure: Number; unit: Participants
Groups:
- All Subjects: Subjects applied both study products in a split-face fashion through week 2. Study products were applied once-daily in the evening.
Arm/Group | All Subjects
Number analyzed (Participants) | 47
Participants
  Week 1, Epiduo Gel, n=47 | 15
  Week 1, Clindoxyl Gel, n=47 | 30
  Week 1, Both Treatments Equally, n=47 | 2
  Week 2, Epiduo Gel, n=46 | 16
  Week 2, Clindoxyl Gel, n=46 | 29
  Week 2, Both Treatments Equally, n=46 | 1

32. Secondary Outcome: Product Acceptability and Preference Questionnaire - Comparison of Study Products Used in the Past at Week 8
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 1, More Satisfied; 2, Somewhat More Satisfied; 3, Neither Satisfied or Dissatisfied; 4, Somewhat More Dissatisfied; 5, More Dissatisfied.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 1.63 (1.08)

33. Secondary Outcome: Product Acceptability and Preference Questionnaire - Decrease of Acne Breakouts by Study Products at Weeks 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint using the following scale: 1, Highly Favorable; 2, Favorable; 3, Neutral; 4, Unfavorable; 5, Uncomfortable.
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 1.87 (0.68) | 2.04 (0.78)
  Week 2 | 1.85 (0.84) | 2.00 (0.70)

34. Secondary Outcome: Product Acceptability and Preference Questionnaire - Decrease of Acne Breakouts by Study Products at Week 8
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 1, Highly Favorable; 2, Favorable; 3, Neutral; 4, Unfavorable; 5, More Dissatisfied.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Clindoxyl Gel: Subjects applied Clindoxyl gel to the entire face once-daily in the evening.
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 1.53 (0.65)

35. Secondary Outcome: Product Acceptability and Preference Questionnaire - Compliance at Weeks 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint using the following scale: 0, Not Compliant at all; 1, Mostly Compliant; 2, Very Compliant.
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 1.91 (0.28) | 1.91 (0.28)
  Week 2 | 1.85 (0.42) | 1.85 (0.42)

36. Secondary Outcome: Product Acceptability and Preference Questionnaire - Compliance at Week 8
Description: Product Acceptability and Preference Questionnaire were completed by the subject at week 8 by answering Yes or No to the following question: Did you use the product every day?. When only one product was applied to the face, subjects were asked to rate their compliance by answering the aforementioned question, rather than rating compliance on a 0-2 scale.
Time Frame: Week 8
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Participants
  Yes | 43
  No | 3

37. Secondary Outcome: Product Acceptability and Preference Questionnaire - Feeling of Hydrated and Moisturized Skin at Weeks 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint by answering Yes or No to the following question: Did you feel that your skin was hydrated and moisturized while you were on your study product?
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Participants
  Week 1 - Yes | 16 | 12
  Week 1 - No | 31 | 35
  Week 2 - Yes | 14 | 11
  Week 2 - No | 32 | 35

38. Secondary Outcome: Product Acceptability and Preference Questionnaire - Feeling of Hydrated and Moisturized Skin at Week 8
Description: as for outcome 37
Time Frame: Week 8
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Participants
  Yes | 28
  No | 18

39. Secondary Outcome: Product Acceptability and Preference Questionnaire - Use of Study Product if Choice to Continue Acne Treatment at Week 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint by answering Yes or No to the following question: If you were to choose to continue treatment for your acne, would you use the study product?
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Participants
  Week 1 - Yes | 44 | 26
  Week 1 - No | 3 | 21
  Week 2 - Yes | 39 | 32
  Week 2 - No | 7 | 14

40. Secondary Outcome: Product Acceptability and Preference Questionnaire - Use of Study Product if Choice to Continue Acne Treatment at Week 8
Description: Product Acceptability and Preference Questionnaire were completed by the subject at 8 week timepoint by answering Yes or No to the following question: If you were to choose to continue treatment for your acne, would you use the study product?
Time Frame: Week 8
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Participants
  Yes | 41
  No | 5

41. Secondary Outcome: Product Acceptability and Preference Questionnaire - Ease of Use Wtih Make-Up at Weeks 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint using the following scale: 0, Not Applicable; 1, Very Easy; 2, Easy; 3, Neutral; 4, Difficult; 5, Very Difficult.
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 2.23 (1.24) | 2.31 (1.38)
  Week 2 | 1.75 (0.93) | 1.75 (0.93)

42. Secondary Outcome: Product Acceptability and Preference Questionnaire - Ease of Use With Make-Up at Week 8
Description: as for outcome 41
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 1.69 (0.87)

43. Secondary Outcome: Product Acceptability and Preference Questionnaire - Overall Satisfaction of Study Product at Weeks 1 and 2
Description: Product Acceptability and Preference Questionnaire were completed by the subject at each timepoint using the following scale: 1, Very Satisfied; 2, Satisfied; 3, Neutral; 4, Unsatisfied; 5, Very Unsatisfied.
Time Frame: Weeks 1 and 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel | Epiduo Gel
Number analyzed (Participants) | 48 | 48
Units on a scale
  Week 1 | 2.09 (0.69) | 2.23 (0.87)
  Week 2 | 1.76 (0.77) | 1.98 (0.68)

44. Secondary Outcome: Product Acceptability and Preference Questionnaire - Overall Satisfaction of Study Product at Week 8
Description: as for outcome 43
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindoxyl Gel
Number analyzed (Participants) | 48
Units on a scale | 1.61 (0.98)

ADVERSE EVENTS:
Time Frame: Baseline through Week 8.
Description: Any study product-related AEs ongoing at the end of the treatment period will be followed until they resolve, the condition stabilizes, the events are otherwise explained, or the subject is lost to follow-up. In addition, all SAEs will be followed until resolution as previously stated for study product-related AEs.
Arm/Group | Clindoxyl and Epiduo Gels
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 44/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clindoxyl and Epiduo Gels (N=48)
Application site irritation (Skin and subcutaneous tissue disorders) | 36 (36)
Application site dryness (Skin and subcutaneous tissue disorders) | 19 (19)
Application site pruritus (Skin and subcutaneous tissue disorders) | 11 (11)
Application site exfoliation (Skin and subcutaneous tissue disorders) | 10 (10)
Drug intolerance (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Investigator wishes to make any such publication or presentation, the Investigator must first submit such publication or presentation to Stiefel for review at least thirty (30) days prior to the date on which such publication or presentation is proposed to be made.